CLINICAL TRIAL: NCT00442767
Title: Reducing Postprandial Hyperglycemia With Adjuvant Premeal Pramlintide and Postmeal Insulin in Children With Type 1 Diabetes Mellitus.
Brief Title: Post-meal Insulin Dosing With Adjuvant Pre-meal Pramlintide in Children With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Rubina Heptulla, Principal Investigator, Montefiore Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-18629; GCRC protocol #:0954
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: pediatric; juvenile; diabetes mellitus; Pediatric type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin; Insulin Aspart; Insulin Lispro; pramlintide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapid acting Insulin therapy - before meal (Active Comparator): Insulin therapy was continued as per prescribed home regimen without pramlintide. Subjects self-administered a rapid-acting insulin analog (aspart or lispro) bolus based on their individual insulin: carbohydrate ratio, before meal
  Interventions: Drug: Insulin
- Pre-meal Pramlintide and Post-meal Insulin therapy (Experimental): 30mcg of pramlintide was administered subcutaneously immediately prior to the meal and insulin was given 15 minutes after the meal. The dose of insulin was reduced by 20%.
  Interventions: Drug: Pramlintide + Insulin

INTERVENTIONS:
Drug: Insulin — Insulin therapy was continued as per prescribed home regimen without pramlintide. Subjects self-administered a rapid-acting insulin analog (aspart or lispro) bolus based on their individual insulin: carbohydrate ratio, before meal.
  Other Names: aspart or lispro
  Arms: Rapid acting Insulin therapy - before meal
Drug: Pramlintide + Insulin — 30mcg of pramlintide was administered subcutaneously immediately prior to the meal and insulin was given 15 minutes after the meal. The dose of insulin was reduced by 20%.
  Other Names: Pramlintide Acetate
  Arms: Pre-meal Pramlintide and Post-meal Insulin therapy

SUMMARY:
The primary objective of this study is to examine the effect of pramlintide given pre-meal and insulin given just after a meal vs. standard therapy of pre-meal insulin on post-prandial glucose excursions.

The secondary objective is to examine the effect of pramlintide and insulin on glucagon suppression in type 1 diabetes.

DETAILED DESCRIPTION:
Following approval by the Institutional Review Board at Baylor College of Medicine 8 adolescents (6 males, 2 females) with type 1 diabetes were recruited to the open-labeled, non-randomized, crossover study. Two male subjects were African American; the remaining subjects were all Caucasian. Six subjects were on insulin pump therapy, and the two on insulin glargine, self-administered at -90minutes. Subjects had their last meal before 12 midnight, and stayed at our research center from 7AM until completion of the study at 2PM. Study A was done before study B.

Basal insulin doses of the subjects were kept constant through studies A and B. No subject was prescribed pramlintide any time in the past prior to participation in this study.

Study A:Insulin therapy was continued as per prescribed home regimen without pramlintide. Subjects self-administered a rapid-acting insulin analog (aspart or lispro) bolus based on their individual insulin: carbohydrate ratio, following which they received 12oz (591ml) of Boost High Protein drink (360 calories, 50gms carbohydrate, 12 gms fat) at 9AM (0 minutes). The Boost was consumed in 5 - 7 minutes. Blood samples were collected for the analysis of blood glucose (BG) levels at -60, -30, -10, and 0 minutes, and every 10 minutes thereafter for the first hour, every 20 minutes for the second hour, and every 30 minutes until the study ended. Blood samples were also collected throughout the study at multiple time points for the analysis of insulin and glucagon levels. Subjects were provided with lunch at 2PM, and discharged.

Study B:The study protocol was identical to study A except 30mcg of pramlintide was administered subcutaneously immediately prior to drinking the Boost at 9AM, and no insulin was given before the meal but was given 15 minutes after the meal (9:15AM) and the dose was reduced by 20%. Study B was conducted within 3 to 4 weeks of study A.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes only
* Diagnosed with T1DM for at least 1 year
* HbA1C less than or equal to 8.5%
* Currently treated using insulin glargine with or without Humalog/ Novolog or on the insulin pump
* Hemoglobin equal to or greater than 12mg/dL
* Otherwise healthy, EXCEPT for T1DM and treated hypothyroidism
* Negative pregnancy test, in the case of females

Exclusion Criteria:

* Lack of supportive family
* Evidence or history of chemical abuse
* BMI (body mass index) greater than the 90th percentile OR less than the 10th percentile for age
* Patient who is poorly compliant with current insulin management and/or Prescribed self blood glucose monitoring
* Patient who experiences recurrent severe hypoglycemia episodes (requiring assistance/ hospitalizations) in the past 6 months
* Have hypoglycemia unawareness
* Have a confirmed diagnosis of gastroparesis, and/ or require medications that stimulate gastrointestinal motility
* Pregnant or lactating patients, or patients planning on becoming pregnant

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubina A Heptulla, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] Hassan K, Heptulla RA. Reducing postprandial hyperglycemia with adjuvant premeal pramlintide and postmeal insulin in children with type 1 diabetes mellitus. Pediatr Diabetes. 2009 Jun;10(4):264-8. doi: 10.1111/j.1399-5448.2008.00490.x. Epub 2008 Dec 18. PMID 19140902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight study subjects were screened and all subjects completed both study visits.
Groups:
- Insulin Therapy / Pramlintide + Insulin Therapy: Rapid acting Insulin therapy - before meal: Insulin therapy was continued as per prescribed home regimen without pramlintide. Subjects self-administered a rapid-acting insulin analog (aspart or lispro) bolus based on their individual insulin: carbohydrate ratio, before meal.
  Pre-meal Pramlintide and Post-meal Insulin therapy: 30mcg of pramlintide was administered subcutaneously immediately prior to the meal and insulin was given 15 minutes after the meal. The dose of insulin was reduced by 20%.
Period: Overall Study
Arm/Group | Insulin Therapy / Pramlintide + Insulin Therapy
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Insulin Therpy / Pramlintide + Insulin Therapy: Rapid acting Insulin therapy - before meal: Insulin therapy was continued as per prescribed home regimen without pramlintide. Subjects self-administered a rapid-acting insulin analog (aspart or lispro) bolus based on their individual insulin: carbohydrate ratio, before meal.
  Pre-meal Pramlintide and Post-meal Insulin therapy: 30mcg of pramlintide was administered subcutaneously immediately prior to the meal and insulin was given 15 minutes after the meal. The dose of insulin was reduced by 20%.
Arm/Group | Insulin Therpy / Pramlintide + Insulin Therapy
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.2 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Assess the Mean Area Under the Curve (AUC) for Blood Glucose Concentration in Subjects Treated With Pramlintide + Insulin, Compared to Insulin Alone
Description: Blood glucose concentration in terms of mean AUC (0 to 240 minutes) was determined in subjects treated with Pramlintide + Insulin vs. Insulin alone
Time Frame: 0 to 240 minutes post-dose
Measure: Mean (Standard Error); unit: mmol*L/min
Groups:
- Rapid Acting Insulin Therapy - Before Meal: Rapid acting Insulin therapy - before meal: Insulin therapy was continued as per prescribed home regimen without pramlintide. Subjects self-administered a rapid-acting insulin analog (aspart or lispro) bolus based on their individual insulin: carbohydrate ratio, before meal.
- Pre-meal Pramlintide and Post-meal Insulin Therapy: Pre-meal Pramlintide and Post-meal Insulin therapy: 30mcg of pramlintide was administered subcutaneously immediately prior to the meal and insulin was given 15 minutes after the meal. The dose of insulin was reduced by 20%.
Arm/Group | Rapid Acting Insulin Therapy - Before Meal | Pre-meal Pramlintide and Post-meal Insulin Therapy
Number analyzed (Participants) | 8 | 8
mmol*L/min | 205 (116) | 993 (141)

2. Secondary Outcome: Measure of Glucagon Concentration in Subjects Treated With Pramlintide + Insulin, Compared to Insulin Alone.
Description: Glucagon concentration in terms of mean AUC (0 to 120 minutes) was determined in subjects treated with Pramlintide + Insulin vs. Insulin alone
Time Frame: 0 to 120 minutes post-dose
Measure: Mean (Standard Error); unit: ng*L/min
Arm/Group | Rapid Acting Insulin Therapy - Before Meal | Pre-meal Pramlintide and Post-meal Insulin Therapy
Number analyzed (Participants) | 8 | 8
ng*L/min | 6060 (459) | 7575 (479)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Insulin Therapy: Rapid acting Insulin therapy - before meal: Insulin therapy was continued as per prescribed home regimen without pramlintide. Subjects self-administered a rapid-acting insulin analog (aspart or lispro) bolus based on their individual insulin: carbohydrate ratio, before meal.
- Pramlintide + Insulin Therapy: Pre-meal Pramlintide and Post-meal Insulin therapy: 30mcg of pramlintide was administered subcutaneously immediately prior to the meal and insulin was given 15 minutes after the meal. The dose of insulin was reduced by 20%.
Arm/Group | Insulin Therapy | Pramlintide + Insulin Therapy
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No